## Title page

| _ | ٠ | | ı | | |
|---|---|---|---|---|---|
| | ı | t | ı | Δ | • |
| • | ı | L | ı | C | • |

Mesalazine in the Treatment of Hidradenitis Suppurativa: a case series

Date:

August 29, 2024

## Study Protocol:

We performed clinical, laboratory tests and ultrasound evaluations to confirm HS lesions at baseline as well as in the follow-up visits. The patients were divided into mild to moderate group (Hurley stage I, II) and severe group(Hurley stage III). Their baseline score on the the IHS4 and DLQI scales before and after starting the treatment were compared. We also registered the number of patients who achieved HiSCR.

## Statistical Analysis Plan:

All the collected data were integrated, and SPSS 26 statistical software was used for data analysis. After normality test, the measurement data were described by mean  $\pm$  standard deviation if they met normal distribution. Those who did not fit were described by median (upper quartile, lower quartile).

The measurement data were tested for normality, and if they fit normal distribution, analysis of variance was performed. If the variance is homogeneous, the t test is used, otherwise the approximate t test is used. If the data does not conform to a normal distribution, the rank sum test is used. For rank data, ordered regression analysis and independent sample rank sum test were used. In statistical analysis, a P-value less than 0.05 indicates a statistical difference. A P-value of less than 0.01 indicates a statistically significant difference.